CLINICAL TRIAL: NCT01283165
Title: Analysis on the Burden of Helminths-plasmodium Polyparasitism, Impact on Anaemia and Effects of Integrated School Based Parasite Control and Health Education in Zimbabwe
Brief Title: Worm Infestation and Child Health in Zimbabwe
Acronym: Zimworms
Status: Completed | Type: Observational
Sponsor: University of Zimbabwe (Other)
Collaborators: National Institute of Health Research, Zimbabwe (Other Government)
Responsible Party: Takafira Mduluza Professor, Biochemistry Department, University of Zimbabwe
Other Study IDs: ZimWorm
Record Dates: First submitted 2011-01-24; First posted 2011-01-25 (Estimated); Last update posted 2011-11-10 (Estimated); Status verified 2003-01

CONDITIONS: Integrated Control of Malaria and Polyparasitism
Keywords: health education; Polyparasitism; school based deworming program; integrated control of parasites
MeSH Terms: conditions — Health Education

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- health education: This was an intervention follow up Knowledge Attitude and Practice study that investigated the distribution of polyparasitism with schistosomiasis, STHs and P. falciparum among primary schoolchildren.
  Interventions: Behavioral: Health education intervention

INTERVENTIONS:
Behavioral: Health education intervention — Health education was conducted in two ways. (1) Teachers were taught how to use the flip chart that contained health education material about parasites. The lessons were done during free periods as this intervention had not been formally fitted into the school syllabus. (2) The research team provided health education to school children. Focus group discussions were conducted by the research team with school children all assembled outside their classes. Health education leaflets were distributed to all school children at the school. Children were asked to share the health information with their friends and families.
  Other Names: Knowledge Attitude and Practice intervention

SUMMARY:
The main objective of the project was to determine the effect of integrated school based deworming and health education on prevalence and morbidity due to co-infection infection with schistosomiasis, STHs and malaria among primary school age children living in rural and farming areas in Zimbabwe

There is need for regular school based de-worming and health education programs for the helminths-Plasmodium co-infections in primary schoolchildren living in rural and commercial farming areas in Zimbabwe

DETAILED DESCRIPTION:
Schistosomiasis is one of the major communicable diseases of public health and socio-economic importance in the developing world. More than 600 million people are at risk of infection with schistosomiasis, 207 million are infected and 120 million are suffering from severe morbidity due to schistosomiasis. Soil transmitted helminths (hookworms, Trichuris trichura and Ascaris lumbricoides) infect more than 2 billion people with children being the most at risk age group. Common clinical outcomes of soil transmitted helminths (STHs) include anaemia, impaired physical development, cognition and malnutrition area especially in primary school children. Global estimates indicate 243 million cases of malaria worldwide of which (85%) were reported in African region only. It accounted for an estimated 863 000 deaths in 2008, of which 89% occurred in the Africa alone.

The high prevalence of schistosomiasis, STHs and malaria and the striking similarity of the conditions that favour their survival, reproduction and transmission that include poverty, lack of preventive measures, health care, safe water and sanitary facilities, and the similarity in temperatures conditions, make polyparasitism from these parasites a "norm that an exception" in tropical and sub-tropical areas. Separate studies have shown endemicity of schistosomiasis, STHs and malaria in Zimbabwe and all these studies have demonstrated high prevalence of schistosomiasis, STHs and malaria among primary schoolchildren. Though only single parasite were investigated in separate studies, results from previous studies indicate geographic overlap of helminths and Plasmodium and thus polyparasitism especially in primary schoolchildren. However data is scarce on extend of polyparasitism with schistosomiasis, STHs and Plasmodium malaria in Zimbabwe and else where. Delineation of areas co-endemic for helminthiasis and malaria and the knowledge of the proportion of the population with co-infections is a first step in allocating limited public health resources for integrated control programmes. Using parasitological methods this study sought to determine the distribution of polyparasitism in primary schoolchildren living in rural and commercial farming areas in Zimbabwe.

Prevalence of anaemia among children under 5 years of age in Zimbabwe is 58% (range 55.4%-63.1%) and it is 38% (range 30.7%-47.5%) for women. However the prevalence of anaemia in primary school age children (5-15 years) is not reported. Neither is there a report on the etiology of anaemia in this age group. Data is also lacking on the contribution of STHs, schistosomiasis and Plasmodium falciparum on the reported anaemia prevalence in Zimbabwe although they are major contributors to this disease. There is also a paucity of evidence on the impact of polyparasitism with helminths and Plasmodium on anaemia especially among the most susceptible primary schoolchildren in the developing world including Zimbabwe. These gaps derail policy decisions on appropriate integrated control strategies that should be based on scientific evidence from field studies. The impact of polyparasitism on anaemia among primary schoolchildren living in the commercial farming area was determined in this study.

The growing interest for the global control of polyparasitism by combining different interventions is economically considered cost effective and the global attention is focused on this strategy. However a number of operational research questions including the choice of different integrated control strategies, timing of treatment cycles, feasibility of implementation and impact on prevalence of polyparasitism, and anaemia requires evaluation before rolling out large scale control programmes. A longitudinal study was conducted to investigate the impact of combined regular school based treatment and delayed treatment of parasitic diseases on polyparasitism and anaemia.

Zimbabwe is among WHO member states that have placed control of schistosomiasis, malaria and STHs high on the agenda. Wide spread use of Praziquantel will be inevitable. However whilst global use of Praziquantel is scaling up, there is also a growing concern in the use of this single drug for treatment of a disease affecting more than 200 million people especially in the wake of low cure rates reported in Senegal and Egypt. Consequently recommendations for continued monitoring for Praziquantel resistance under the pressure of wide spread use of the drug have been made. Current data is lacking on the efficacy of Praziquantel in treatment of schistosomiasis in Zimbabwean population. Praziquantel drug efficacy was determined in this study in order to advice health managers on the implications of mass drug administration that is pending as Zimbabwe prepares from mass treatment using the school based approach.

The World Health Organization recommends that any large scale control programme should be preceded by a baseline survey in order to monitor and evaluate control strategies during and after implementation. For the control of helminthiasis, conducting the baseline survey in grade three children (8-10years) is recommended since they harbour the highest prevalence and intensity of infection in the community and can be followed up to at least two years to monitor and evaluate effectiveness of any control strategy implemented. Thus the prevalence of helminths in this age group can be used as an index for assessing community prevalence. However data on Knowledge attitudes and practice (KAP) of grade three children in relation to schistosomiasis, STHs and malaria is lacking. The impact of school health education on behaviour modification of the school children towards prevention of helminthiasis and malaria in Zimbabwe is also scarce. A follow up KAP study was conducted in grade three children before and after school based health education integrated with treatment.

ELIGIBILITY:
Inclusion Criteria:

* all school children at the primary schools

Exclusion Criteria:

* Very sick with known TB or HIV infection

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Primary school going children living in rural and commercial farming areas
Sampling Method: Non-Probability Sample
Enrollment: 1303 (Actual)
Dates: Start 2003-04; Primary Completion 2006-06 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
This study was conducted to determine the prevalence of polyparasitism among primary school children living in rural and commercial farming areas in Zimbabwe. | 3 years
  This study was conducted to determine the prevalence of polyparasitism, the impact of polyparasitism on anaemia, the effect of combined school based treatment for STHs, schistosomiasis, health education and prompt malaria treatment on anaemia and prevalence of polyparasitism in primary school children.

SECONDARY OUTCOMES:
Impact of school based parasite treatment and health education intervention. | 3 years
  To determine the impact of combined school based deworming and prompt malaria treatment on prevalence of helminths-Plasmodium co-infections, anaemia and severity of anaemia among primary schoolchildren in rural and commercial farming areas in Zimbabwe. Combined school based parasite treatment were performed at baseline and at each follow up survey. Sustained prompt malaria treatment was performed throughout the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Takafira Mduluza, PhD, Principal Investigator — University of Zimbabwe
Locations (1):
- Biochemistry Department University of Zimbabwe, Harare, Zimbabwe

REFERENCES:
- [Result] Midzi N, Mtapuri-Zinyowera S, Mapingure MP, Sangweme D, Chirehwa MT, Brouwer KC, Mudzori J, Hlerema G, Mutapi F, Kumar N, Mduluza T. Consequences of polyparasitism on anaemia among primary school children in Zimbabwe. Acta Trop. 2010 Jul-Aug;115(1-2):103-11. doi: 10.1016/j.actatropica.2010.02.010. Epub 2010 Feb 20. PMID 20175980
- [Result] Midzi N, Sangweme D, Zinyowera S, Mapingure MP, Brouwer KC, Munatsi A, Mutapi F, Mudzori J, Kumar N, Woelk G, Mduluza T. The burden of polyparasitism among primary schoolchildren in rural and farming areas in Zimbabwe. Trans R Soc Trop Med Hyg. 2008 Oct;102(10):1039-45. doi: 10.1016/j.trstmh.2008.05.024. Epub 2008 Jul 24. PMID 18656215
- [Result] Midzi N, Sangweme D, Zinyowera S, Mapingure MP, Brouwer KC, Kumar N, Mutapi F, Woelk G, Mduluza T. Efficacy and side effects of praziquantel treatment against Schistosoma haematobium infection among primary school children in Zimbabwe. Trans R Soc Trop Med Hyg. 2008 Aug;102(8):759-66. doi: 10.1016/j.trstmh.2008.03.010. Epub 2008 May 16. PMID 18486169
- See also: Medical Research Council of Zimbabwe — http://www.mrcz.org.zw